CLINICAL TRIAL: NCT01654926
Title: Feasibility Assessment of the Aquadex FlexFlowTM Ultrafiltration System in Treating Non Hospitalized Heart Failure Patients in Dedicated Heart Failure Centers
Status: Completed | Type: Observational
Sponsor: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Dr. Ofer Amir, Head of the Lin Heart Failure Center, Clalit Health Services
Other Study IDs: UF-HF-1
Record Dates: First submitted 2012-07-29; First posted 2012-08-01 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Heart Failure
Keywords: Feasibility of using the FlexFlowTM ultrafiltration pump in a non hospital environment
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Failure patients
  Interventions: Procedure: blood ultrafiltration

INTERVENTIONS:
Procedure: blood ultrafiltration

SUMMARY:
Ultrafiltration (UF) technology is unique for its ability to extract fluid as an isotonic solution, therefore not causing substantial changes in NaCl concentrations, and the use of peripheral veins makes it feasible to use in out of hospital medical centers, for non compensated Heart Failure (HF) with a low response to diuretics. The use of UF in the United States and Europe in out of hospital HF centers is accepted as daily practice. Therefore the hypothesis of this study is that it is feasible for a professional team to effectively use the UF for short courses on non compensated HF patients with low or no response to Diuretics, in a dedicated out of hospital HF center.

DETAILED DESCRIPTION:
The patients will be treated in the LIN Heart Failure Center and will not include population defined in the Exclusion criteria.

Up to 60 patients will be recruited and each one will undergo up to 30 treatments in time intervals defined by the cardiologist according to the clinical needs throughout the duration of the study.

Inclusion duration of every patient will be terminated at the end of the treatment course. No prevention in adding more treatment courses per patient according to clinical needs upon the cardiologist's decision.

Operating the UF system:

During the treatment course two of the patient's peripheral veins will be cannulated. One will be used to draw blood from, and the other will be used to return the blood back in to the patient.

The patient will be administered with Heparin IV, or Clexane SC with an ACT target of 180-200 that will be monitored every 4-6 hours.

Fluid removal rate will be according to the cardiologists discretion and will not exceed 500 ml/hour Patient monitoring - Pulse and BP will be recorded at baseline, after 10 minutes for treatment onset and every 1 hour.

ELIGIBILITY:
Inclusion Criteria:

HF patients with peripheral or pulmonic fluid retention, with little or no response to Diuretics as defined by the referring cardiologist

Exclusion Criteria:

1. Age < 18 years
2. Patient does not fully comprehend the Essence of the study and can not sign the informed consent.
3. Patient is participating in a drug or any other treatment study (no prevention to include patients participating in studies of non invasive monitoring technologies.
4. Presence of Acute MI
5. CR base values > 3mg/dl
6. Hemodynamic instability requiring Inotropic agents
7. HT base values > 45%
8. Known pregnancy
9. Presence of contraindication to anticoagulants
10. Post heart transplant or cardiac assist device implantation

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HF patients
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Feasibility Assessment of the Aquadex FlexFlowTM Ultrafiltration System in Treating Non-Hospitalized Heart Failure Patients in Dedicated Heart Failure Centers | 12 months
  The propose of the study is to observe the administrative needs of performing the treatment at our specific out-patient clinic. Of note the treatment is already approved including the indication and the place we are doing it so we merely aim to look at administrative and logistic that need to be done.

CONTACTS AND LOCATIONS:
Locations (1):
- Lin Clinic, Haifa, Israel